CLINICAL TRIAL: NCT03917056
Title: Cap-assisted Endoscopic Sclerotherapy for Internal Hemorrhoids and Rectal Prolapse: a Nationwide Multicenter Randomized Controlled Trial
Brief Title: Cap-assisted Endoscopic Sclerotherapy for Internal Hemorrhoids and Rectal Prolapse
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Faming Zhang, Professor, Gastroenterology, The Second Hospital of Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAES-CN-190318
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Internal Hemorrhoid; Rectal Prolapse
Keywords: Cap-assisted endoscopic sclerotherapy; Internal Hemorrhoid; Rectal Prolapse
MeSH Terms: conditions — Rectal Prolapse

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Long needle group (Experimental): Participants were treated with CAES using long needle.
  Interventions: Procedure: Cap-assisted endoscopic sclerotherapy using long needle
- Short needle group (Experimental): Participants were treated with CAES using short needle.
  Interventions: Procedure: Cap-assisted endoscopic sclerotherapy using short needle

INTERVENTIONS:
Procedure: Cap-assisted endoscopic sclerotherapy using long needle — Participants were treated with CAES using long needle.
  Arms: Long needle group
Procedure: Cap-assisted endoscopic sclerotherapy using short needle — Participants were treated with CAES using short needle.
  Arms: Short needle group

SUMMARY:
This clinical trial aims to evaluate the efficacy and safety of long needle and short needle in the treatment of internal hemorrhoids and rectal prolapse through CAES (Cap-assisted endoscopic sclerotherapy).

DETAILED DESCRIPTION:
Traditional endoscopic sclerotherapy for internal hemorrhoids require retroflection of the endoscope. Retroflection of the endoscope has blind areas and affects the precise operation. And, short-needle injection can easily lead to artificial ulcer and secondary bleeding. CAES is a new, minimally invasive endoscopic technique for the treatment of internal hemorrhoids and rectal prolapse. CAES was performed based on the requirement of the cap, endoscope, disposable endoscopic long injection needle, enough insufflated air and sclerosing agent. It can accurately control the injection angle, direction and depth under direct vision, and avoid iatrogenic injury caused by ectopic injection to the greatest possible extent. To investigate the effect of long needle and short needle on the outcome of CAES, participants with internal hemorrhoids and rectal prolapse were randomly assigned to a long needle group and a short needle group using a prospective, randomized, controlled study at multiple centers in China. The efficacy, adverse events and satisfaction of the two groups were observed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with internal hemorrhoids and rectal prolapse, combined with external hemorrhoids or without external hemorrhoids.
2. Patients with bowel preparation.

Exclusion Criteria:

1. History of anoscopic/endoscopic sclerotherapy.
2. Patients with acute thrombotic external hemorrhoids.
3. Patients with serious internal hemorrhoids of grade IV.
4. Patients with anal stenosis, anal fissure, fistula, fecal incontinence, ulcerative colitis, Crohn's disease.
5. Patients with acute diarrhea in the past 24 hours.
6. Hypertensive patients with uncontrolled blood pressure, patients with cerebrovascular accident and obvious bleeding tendency, pregnant women, mental disorders and decompensated cirrhosis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2019-06-24 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-27 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | 24 weeks
  Recurrence rate defined as the proportion of patients with recurrent hemorrhoids at 24 weeks post-CAES, as derived from patients' self-reported answer. Patients will be considered to have recurrent hemorrhoids when any of the following are recorded: (1)"Unchanged or worse compared with before starting treatment" at 24th week as reported by the patient, or (2) seeking repeat CAES treatment, alternative non-surgical/surgical treatments for internal hemorrhoids within 24weeks (except medication treatment), or (3) presence of any symptoms or events that strongly indicated recurrent hemorrhoids among patients not meeting (1) or (2).

SECONDARY OUTCOMES:
Symptoms of anal bleeding | 1day, 7days, 14days and 24 weeks
  Bleeding is divided into three degrees: 1. No bleeding; 2. 2: occasionally; 3: quite often.
Symptoms of prolapse | 1day, 7days, 14days and 24 weeks
  There are three degrees of prolapse: 1. No prolapse; 2: occasionally; 3: quite often.
Symptoms of anal pain | 1day, 7days, 14days and 24 weeks
  NRS pain digital rating scale was adopted, that is, 0-10 was used to represent different degrees of pain, 0 was painless, and 10 was severe pain. 0 painless, 1-3 mild pain (pain does not affect sleep), 4-6 moderate pain, 7-9 severe pain (inability to fall asleep or waking up during sleep), 10 severe pain.
EQ-5D health scale scores | 24 weeks
  Before CAES and after CAES, EQ-5D health scale scores were performed.
Adverse events and serious adverse events | 1day, 7days, 14days and 24 weeks
  Adverse events included bleeding, anal pain, and dyspnea.Serious adverse events include serious complications directly or indirectly related to the operation, such as death, bleeding, perforation, etc.
Satisfaction degree | 24 weeks
  Number of satisfied participants
Symptom severity score | 1day and 24 weeks
  five questions about hemorrhoidal symptoms (anal pain, prolapse, itching, soiling, and blood loss) will be self-assessed by patients by answering how often each symptom was encountered (never, sometimes, weekly, or daily). The score is the sum of the points from all five questions, ranging from 0 to 15 points, where an increase in number is an increase in symptom.

CONTACTS AND LOCATIONS:
Overall Officials: Faming Zhang, MD,PhD, Principal Investigator — The Second Hospital of Nanjing Medical University
Locations (1):
- Fmt-Dt-N-27/1350, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Zhang T, Xu LJ, Xiang J, He Z, Peng ZY, Huang GM, Ji GZ, Zhang FM. Cap-assisted endoscopic sclerotherapy for hemorrhoids: Methods, feasibility and efficacy. World J Gastrointest Endosc. 2015 Dec 25;7(19):1334-40. doi: 10.4253/wjge.v7.i19.1334. PMID 26722615
- [Background] Tomiki Y, Ono S, Aoki J, Takahashi R, Sakamoto K. Endoscopic sclerotherapy with aluminum potassium sulfate and tannic acid for internal hemorrhoids. Endoscopy. 2014;46 Suppl 1 UCTN:E114. doi: 10.1055/s-0034-1364884. Epub 2014 Mar 27. No abstract available. PMID 24676816
- [Derived] Wu X, Wen Q, Cui B, Liu Y, Zhong M, Yuan Y, Wu L, Zhang X, Hu Y, Lv M, Wu Q, He S, Jin Y, Tian S, Wan R, Wang X, Xu L, Bai J, Huang G, Ji G, Zhang F. Cap-assisted endoscopic sclerotherapy for internal hemorrhoids: technique protocol and study design for a multi-center randomized controlled trial. Ther Adv Gastrointest Endosc. 2020 Jun 5;13:2631774520925636. doi: 10.1177/2631774520925636. eCollection 2020 Jan-Dec. PMID 32551439